CLINICAL TRIAL: NCT05884879
Title: Assessment of Listening Effort in Tinnitus Patients
Brief Title: Listening Effort in Tinnitus Patients
Acronym: ALERT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 301849
Record Dates: First submitted 2023-04-28; First posted 2023-06-01 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2023-05

CONDITIONS: Listening Effort; Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tinnitus group: * Adults, i.e. 18-69 year old;
  * Pure tone average <35 dB HL (0.5, 1, 2, 4 kHz);
  * Proficient and native speaker of Dutch language;
  * Severe unilateral or bilateral tinnitus disorder (TQ > 46).
- Control group: * Adults, i.e. 18-69 year old;
  * Pure tone average <35 dB HL (0.5, 1, 2, 4 kHz);
  * Proficient and native speaker of Dutch language;
  * No tinnitus.
  Interventions: Behavioral: Tinnitus simulation

INTERVENTIONS:
Behavioral: Tinnitus simulation — The control group will perform speech perception tests and listening effort tests in the absence and presence of a simulated tinnitus percept using a bone vibrator.
  Groups: Control group

SUMMARY:
About 5-15% of the general population experience a chronic ringing, buzzing, hissing or roaring sound in one or two ears, without any external source. This so-called tinnitus can be present in people with normal hearing, but often coexists with hearing loss. Most people suffering from tinnitus can cope with it, however a minority experiences emotional distress or cognitive dysfunction as a result of the tinnitus, called tinnitus disorder. People suffering from tinnitus disorder regularly complain about an increased experienced effort when listening to speech or other sounds in daily life situations. As this has never been proven scientifically, the investigators aim to evaluate the effect of the tinnitus percept and tinnitus disorder on experienced listening effort by comparing listening effort between a population with tinnitus disorder and a population without tinnitus.

ELIGIBILITY:
Inclusion Criteria:

* Young adults, i.e. 18-69 year old;
* Pure tone average <35 dB HL (0.5, 1, 2, 4 kHz);
* Proficient and native speaker of Dutch language;
* TINNITUS GROUP: Severe unilateral or bilateral tinnitus disorder (TQ > 46).
* CONTROL GROUP: No tinnitus.

Exclusion Criteria:

* Significant asymmetric hearing loss: |PTAright - PTAleft| > 15 dB (PTA = pure tone average of 500, 1000, 2000 and 4000 Hz);
* Significant loss of vision (text on screen at 70 cm should be readable);
* Frequent user of any of the following devices: Hearing Aid, Bone Conduction Device, Cochlear Implant, Tinnitus Masker;
* Additional mental or physical disabilities that may prevent active participation and testing as per protocol.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: TINNITUS GROUP:
  Tinnitus patients visiting the Audiological Centre of Maastricht UMC+, Adelante Zorggroep Hoensbroek and Blerick, Libra Eindhoven, Kentalis Eindhoven, Den Bosch and Nijmegen.
  CONTROL GROUP:
  General population visiting the Maastricht UMC+.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Listening effort | 1 day
  Subjective listening effort as a function of the speech reception threshold (SRT)

SECONDARY OUTCOMES:
Listening effort predictability of tinnitus related questionnaire: TQ | 1 day
  Relative importance of sub scales of tinnitus related questionnaires for predicting the amount of listening effort in tinnitus patients:
  Tinnitus Questionnaire (score 0-84, higher score = more tinnitus disorder)
Listening effort predictability of tinnitus related questionnaire: TFI | 1 day
  Relative importance of sub scales of tinnitus related questionnaires for predicting the amount of listening effort in tinnitus patients:
  Tinnitus Functional Index (score 0-100, higher score = more negative impact of tinnitus)
Listening effort predictability of tinnitus related questionnaire: HADS | 1 day
  Relative importance of sub scales of tinnitus related questionnaires for predicting the amount of listening effort in tinnitus patients:
  Hospital Anxiety and Depression Scale (score 0-21, higher score = more anxiety and/or depression)

CONTACTS AND LOCATIONS:
Overall Officials: Erwin LJ George, MPE PhD, Principal Investigator — Maastricht UMC
Locations (1):
- Maastricht UMC+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No